CLINICAL TRIAL: NCT00240955
Title: Efficacy and Safety of Two Immunosuppressive Regimens Mycophenolate Sodium (EC-MPS) With Short-term Steroid Use or Free of Steroids Compared With a Regimen of EC-MPS With Standard Steroids in de Novo Kidney Recipients
Brief Title: Extension Study of Enteric-coated Mycophenolate Sodium With Short-term or no Steroid Use Compared With Enteric-coated Mycophenolate Sodium With Standard Steroid Therapy in de Novo Kidney Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CERL080A2404E1
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Renal Transplantation
Keywords: Renal/Kidney, Transplantation, steroids, EC-MPS

INTERVENTIONS:
Drug: Enteric-coated Mycophenolate sodium (EC-MPS)

SUMMARY:
The objective of this study is to assess the long-term safety and tolerability of EC-MPS on the patients who completed the core study and wish to continue treatment on EC-MPS.

ELIGIBILITY:
Inclusion Criteria/ Exclusion Criteria

* All patients who completed the core study and who are still receiving the EC-MPS and wish continue treatment with EC-MPS and from whom written informed consent has been obtained

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2004-03; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of enteric-coated mycophenolate sodium based on adverse event (AE) reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis